CLINICAL TRIAL: NCT00494143
Title: Metabolic Cost Savings for Transtibial Amputees Walking With the CESR Foot
Brief Title: Metabolic Cost Savings for Transtibial Amputees Wearing the Controlled Energy Storage and Return (CESR) Foot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4372-R
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Transtibial Amputation
Keywords: Amputee; Economy; Efficiency; Foot; Gait; Kinematics; Kinetics; Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional Prosthetic foot (Active Comparator): A conventional prosthetic foot that has limited energy storage and return capabilities. It is standardized and used by all subjects in the study.
  Interventions: Device: typical prosthetic foot
- Prescribed Prosthetic foot (Active Comparator): the Prosthetic foot that the subject had prescribed for them by their clinical providers and was worn prior to study initiation
  Interventions: Device: standardized prosthetic foot
- CESR foot (Experimental): the experimental CESR, controlled energy storage prosthetic foot
  Interventions: Device: CESR Prosthetic Foot

INTERVENTIONS:
Device: CESR Prosthetic Foot — a novel prosthetic foot that is designed to store energy and release it at a predetermined time in the gait cycle
  Arms: CESR foot
Device: typical prosthetic foot — patients will wear the prosthetic foot that they were prescribed by the care providers in the clinical team
  Arms: Conventional Prosthetic foot
Device: standardized prosthetic foot — a standard foot that has had weights applied to match the mass of the CESR foot
  Arms: Prescribed Prosthetic foot

SUMMARY:
To determine if below-knee amputees will walk with better efficiency wearing a CESR foot which stores energy at heel strike and releases energy releases energy during push-off.

DETAILED DESCRIPTION:
Amputees work harder and have greater oxygen cost during ambulation compared to those without limb loss. Therefore, amputees generally walk slower and tire more easily than intact individuals. The loss of the ankle as a propulsive and supportive joint requires the amputee to perform extra muscular work with the hip, trunk and contralateral limb during ambulation. This increased muscular activity consumes additional metabolic energy and means that amputees have to work harder to walk at the same speed as intact individuals. For some amputees, this extra effort is simply not possible, and their loss of functional ambulation leads to a progressive spiral of disuse, reduced capacity and more disuse. Conversely, greater mobility can lead to greater activity and even more successful return to the workplace. The health consequences for amputees who do not maintain functional ambulation is multifactorial and costly, not only in terms of dollars for the institutions committed to their care, but also for the individuals themselves in terms of decreased quality of life, increased disability and pain. Recent developments have resulted in the design of a novel prosthetic foot that uses the energy from compressive forces during heel contact, stores it throughout midstance and releases it at an optimal instant during push-off in late stance. This unique design, with Controlled Energy Storage and Release (CESR) developed by a team at the University of Michigan, Ann Arbor has been shown to reduce the metabolic cost penalty of prosthetic ambulation (i.e. the increased cost over normal walking) by 50% compared to a standard SACH foot, but as yet only intact individuals wearing an aircast boot equipped with the prosthetic feet have been studied. It is likely that the increased energy savings will also be observed in transtibial amputees. Young, active amputees will soon be entering the VA system following operations in Iraq and Afghanistan, and the energy improvements may benefit this new VA patient population. The CESR foot may also provide substantial metabolic cost savings to older less active amputees currently in the VA system. By improving gait efficiency amputees will be better able to keep up with the demands of functional ambulation, remain more active and postpone many of the debilitating consequences of limited mobility. Therefore we propose to first refine the design of the CESR foot focusing on the energy storage and energy release mechanisms of the CESR foot. Several spring characteristics may prove optimal for certain subjects depending upon weight and walking characteristics. This will be an iterative optimization process with power generation and absorption characteristics of the CESR foot evaluated using computerized gait analysis and the lessons used for further refinement. The second phase will involve a three week wear-testing trial to determine if any improvement in gait economy, reduction in fatigue, improvement in comfort, or increase in the amount of daily walking can be achieved. A validated questionnaire will be utilized to determine each amputee's comfort and fatigue during a three week trial in their conventional foot and with the CESR foot. Step counts will be performed on each individual over the entire 3 week period with both the conventional foot and with the CESR foot. We will collect full body gait kinematics (motion) and kinetics (forces) using our Vicon 612 system, and metabolic measurements using our VmaxST to calculate oxygen cost for 24 transtibial amputees while walking with the CESR foot and their conventional foot. This will permit the calculation of the energy storage and release of the foot by inverse dynamics and calculate the net effect upon metabolic energy cost savings during ambulation at several speeds. If the CESR foot is successful in amputee gait these domains, our next step will be to perform a multi-center study with other VA motion laboratories, and eventually collaborate with Ohio Willow Wood, a prominent prosthetic manufacturer who has expressed an interest in bringing the CESR foot to market.

ELIGIBILITY:
Inclusion Criteria:

* Transtibial Amputees > 1 year walking with prosthesis
* Non-amputee control subjects

Exclusion Criteria:

* Additional musculoskeletal pathology
* Cognitive limitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. Czernieki, MD MS, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

REFERENCES:
- [Result] Segal AD, Zelik KE, Klute GK, Morgenroth DC, Hahn ME, Orendurff MS, Adamczyk PG, Collins SH, Kuo AD, Czerniecki JM. The effects of a controlled energy storage and return prototype prosthetic foot on transtibial amputee ambulation. Hum Mov Sci. 2012 Aug;31(4):918-31. doi: 10.1016/j.humov.2011.08.005. Epub 2011 Nov 17. PMID 22100728
- [Result] Morgenroth DC, Segal AD, Zelik KE, Czerniecki JM, Klute GK, Adamczyk PG, Orendurff MS, Hahn ME, Collins SH, Kuo AD. The effect of prosthetic foot push-off on mechanical loading associated with knee osteoarthritis in lower extremity amputees. Gait Posture. 2011 Oct;34(4):502-7. doi: 10.1016/j.gaitpost.2011.07.001. Epub 2011 Jul 30. PMID 21803584
- [Result] Zelik KE, Collins SH, Adamczyk PG, Segal AD, Klute GK, Morgenroth DC, Hahn ME, Orendurff MS, Czerniecki JM, Kuo AD. Systematic variation of prosthetic foot spring affects center-of-mass mechanics and metabolic cost during walking. IEEE Trans Neural Syst Rehabil Eng. 2011 Aug;19(4):411-9. doi: 10.1109/TNSRE.2011.2159018. Epub 2011 Jun 23. PMID 21708509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited through bulletin board ads and through a local VA amputee clinic. Subjects were included if between the ages of 18 and 80 years, had used a prosthesis for grtr than 2 years, wore the prosthesis grtr than 8 hours per day, did not ambulate with u/e aids and had no falls in the prior 6 mo or known neuro or msk deficits.
Pre-assignment Details: Subjects were provided with suitable acclimatization prior to testing with their initial randomized prosthetic foot type.
Groups:
- Conventional, Prescribed, CESR: this is a randomized arm where the sequence of prosthetic use was their conventional foot, followed by prescribed foot, followed by the CESR foot
- Conventional, CESR, Prescribed: The randomized sequence of prosthetic use in this arm was Conventional foot, followed by CESR foot, followed by Prescribed.
- Prescribed, CESR, Conventional: The randomized sequence of this arm was the Prescribed prosthetic foot, followed by the CESR foot followed by the Conventional prosthetic foot
- Prescribed, Conventional, CESR: This arm included individuals who were randomized to the sequence, Prescribed prosthetic foot, conventional foot, CESR foot
- CESR, Prescribed, Conventional: This arm included the individuals who were randomized to the prosthetic foot sequence, CESR foot followed by Prescribed foot, followed by Conventional foot.
- CESR, Conventional, Prescribed: The individuals in this group were randomized to the prosthetic foot sequence, CESR foot, Conventional foot followed by Prescribed prosthetic foot.
Period: Overall Study
Arm/Group | Conventional, Prescribed, CESR | Conventional, CESR, Prescribed | Prescribed, CESR, Conventional | Prescribed, Conventional, CESR | CESR, Prescribed, Conventional | CESR, Conventional, Prescribed
Started | 1 | 2 | 3 | 0 | 1 | 0
Completed | 1 | 2 | 3 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CESR, Prescribed, Conventional: all subjects were randomized to each of the three interventions
Arm/Group | CESR, Prescribed, Conventional
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 7
stature [Mean (Standard Deviation); unit: meters] — height
  meters | 1.85 (.05)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 80.9 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Oxygen Consumption During Ambulation
Description: VO2 was collected at rest and while walking at a controlled walking speed of 1.14 meters/second for 10 minutes until they reached a steady state for 3 minutes. This was repeated for each foot condition. VO2 at the steady state was recorded in ml/min and were subsequently converted to calories and and then to Watts. The data were then corrected for body weight by dividing by weight in Kg. The gross VO2 in Watts/Kg during walking were then adjusted to net VO2 in Watts/kg by subtracting the resting metabolic rate.
Time Frame: Subjects were oriented to the testing protocol and each prosthetic foot on average 5 days prior to data collection and a acclimatization period of 5-10 minutes with each prosthetic foot prior to data collection
Measure: Mean (Standard Deviation); unit: Watts per kilogram
Groups:
- CESR Experimental Prosthetic Foot: the CESR, controlled energy storage prosthetic foot
  CESR Prosthetic Foot : a novel prosthetic foot that is designed to store energy and release it at a predetermined time in the gait cycle
- Conventional Prosthetic Foot: subjects wearing the conventional prosthetic foot
- Prescribed Prosthetic Foot: subjects wearing the prescribed prosthetic foot
Arm/Group | CESR Experimental Prosthetic Foot | Conventional Prosthetic Foot | Prescribed Prosthetic Foot
Number analyzed (Participants) | 7 | 7 | 7
Watts per kilogram | 3.45 (0.59) | 3.13 (0.33) | 2.97 (0.23)

2. Secondary Outcome: Prosthetic Foot Push Off Peak Power
Description: The biomechanical measurement of the power generated by the prosthetic foot during the push off component of stance phase. The peak power output during the push off component of stance phase was calculated in Joules. It was subsequently standardized for body weight in Kgs. The final units were therefore Joules/Kg.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: joules per kilogram
Groups:
- Conventional Prosthetic Foot: results with the conventional prosthetic foot
- Prescribed Prosthetic Foot: results with prescribed prosthetic foot
Arm/Group | CESR Experimental Prosthetic Foot | Conventional Prosthetic Foot | Prescribed Prosthetic Foot
Number analyzed (Participants) | 7 | 7 | 7
joules per kilogram | 0.27 (0.04) | 0.11 (0.03) | 0.15 (0.04)

3. Secondary Outcome: Peak Intact Knee Loading
Description: The biomechanical measure of the first peak of the knee external adduction moment
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: newton meters per kilogram
Groups:
- Conventional Prosthetic Foot: results while wearing the conventional prosthetic foot
- Prescribed Prosthetic Foot: results while wearing the prescribed prosthetic foot
Arm/Group | CESR Experimental Prosthetic Foot | Conventional Prosthetic Foot | Prescribed Prosthetic Foot
Number analyzed (Participants) | 7 | 7 | 7
newton meters per kilogram | 0.451 (0.144) | 0.608 (0.169) | 0.509 (0.132)

ADVERSE EVENTS:
Groups:
- Arm 3 CESR Prosthetic Foot: subjects randomized to the CESR prosthetic foot
- Arm 1 Conventional Prosthetic Foot: subjects randomized to the conventional prosthetic foot
- Arm 2 Prescribed Prosthetic Foot: subjects randomized to the prescribed prosthetic foot
Arm/Group | Arm 3 CESR Prosthetic Foot | Arm 1 Conventional Prosthetic Foot | Arm 2 Prescribed Prosthetic Foot
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Acclimatization to a prosthetic foot type can alter the measured performance. In this study, subjects were most experienced using their prescribed foot. The CESR foot was also only available in one foot size which can affect gait characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes